CLINICAL TRIAL: NCT02668575
Title: Integrating Supportive Care in Cystic Fibrosis: A Pilot Study
Brief Title: Integrating Supportive Care in Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Principal Investigator, Dio Kavalieratos, PhD, Assistant Professor of Medicine, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB#: PRO14110168
Record Dates: First submitted 2016-01-14; First posted 2016-01-29 (Estimated); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Cystic Fibrosis
Keywords: Pulmonary Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention): Patients randomized to the control arm of this study will continue to receive the standard of high-quality CF care provided to all patients at the UPMC CF Center.
- Supportive Care Intervention (Experimental): Patients randomized to the intervention arm will receive a protocolized supportive care intervention from a palliative care nurse practitioner.
  Interventions: Behavioral: Supportive Care Intervention

INTERVENTIONS:
Behavioral: Supportive Care Intervention — Patients in the intervention arm of the study will see a SC specialist during regularly-scheduled CF clinic visits; per usual care, these visits should occur on a quarterly basis. Using a structured intervention manual, these visits will span 30-60 minutes each. Each visit will have a specific focus, such as: 1) comprehensive palliative care assessment; 2) symptom assessment and self-management; 3) advance care planning; and, 4) coping and resilience. Patients requiring follow up with SC before the next CF appointment will receive telephone follow up or an extra SC visit at the discretion of the SC provider.
  Arms: Supportive Care Intervention

SUMMARY:
Individuals living with cystic fibrosis (CF) commonly report high symptom burden, poor quality of life, and additional psychosocial stressors; these burdens are particularly heightened in advanced stages of the disease. Although supportive care (aka palliative care) has been shown to improve many of these outcomes among patients with illnesses such as cancer, no clinical trials to date have tested the impact of supportive care for patients with CF. The purpose of this pilot randomized clinical trial study is to evaluate the feasibility, acceptability, and perceived effectiveness of an embedded supportive care intervention, whereby a supportive care specialist will be integrated within the usual care experience of patients with advanced CF. The investigators will enroll 50 patients with advanced CF, who will be equally randomized to receive this embedded supportive care intervention or usual care. Secondary measures include: patient quality of life, mood, coping style, satisfaction with care, and symptom burden. This study will provide preliminary data to support the development of a larger, definitive, Phase III randomized clinical trial.

DETAILED DESCRIPTION:
As described above.

ELIGIBILITY:
Inclusion Criteria:

* Ability to comprehend English
* Advanced CF

(Any of the following criteria will be indicative of "Advanced CF")

* Baseline supplemental oxygen requirement
* FEV1 ≤ 50%
* Baseline non-invasive mechanical ventilation requirement
* ≥ 2 hospitalizations in the past 12 months for respiratory complications related to CF

Exclusion Criteria:

* Prisoners
* Females who are pregnant
* Prior receipt of specialist SC services
* Cognitive impairments
* Patients younger than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-03-02 (Actual); Primary Completion 2018-11-29 (Actual); Study Completion 2019-10-07 (Actual)

PRIMARY OUTCOMES:
Feasibility of intervention | Up to 9 months (+/- 4 weeks)
  Measured by: eligibility rate, approach-to-consent rate, approach-to-enroll rate, rate of missed intervention sessions, rate of missing data on patient-reported outcomes.
Acceptability of intervention | Up to 9 months (+/- 4 weeks)
  Measured by: proportion of participants who endorse the intervention as acceptable.
Perceived effectiveness of intervention | Up to 9 months (+/- 4 weeks)
  Measured by: proportion of participants who endorse that they believe the intervention to have been beneficial.
Intervention fidelity | Up to 9 months (+/- 4 weeks)
  Evaluate the fidelity of intervention delivery using structured visit checklists to be completed by the interventionist and research staff.

SECONDARY OUTCOMES:
Patient quality of life: Cystic Fibrosis Questionnaire-Revised (CFQ-R) | Up to 9 months (+/- 4 weeks)
  Change in QOL from baseline as measured by the Cystic Fibrosis Questionnaire-Revised (CFQ-R) at 9 months. Due to the pilot nature of this trial, this measure will not be used to assess the efficacy of the intervention.
Patient mood | Up to 9 months (+/- 4 weeks)
  Change in mood from baseline using the Hospital Anxiety and Depression Scale (HADS), reported at 0, 3, 6, 9 months. Due to the pilot nature of this trial, this measure will not be used to assess the efficacy of the intervention.
Coping style | Up to 9 months (+/- 4 weeks)
  Change in coping style from baseline using the Brief COPE, reported at 0, 3, 6, 9 months. Due to the pilot nature of this trial, this measure will not be used to assess the efficacy of the intervention.
Satisfaction with care | Up to 9 months (+/- 4 weeks)
  Change in satisfaction with care from baseline using the FAMCARE-P13, reported at 0, 3, 6, 9 months. Due to the pilot nature of this trial, this measure will not be used to assess the efficacy of the intervention.
Symptom burden | Up to 9 months (+/- 4 weeks)
  Change in symptom burden from baseline using the Edmonton Symptom Assessment Scale (ESAS), reported at 0, 3, 6, 9 months. Due to the pilot nature of this trial, this measure will not be used to assess the efficacy of the intervention.

OTHER OUTCOMES:
Healthcare utilization | Up to 12 months
  The investigators will evaluate various measures of healthcare utilization, such as: ED visits, unplanned hospitalizations, and healthcare expenditures.

CONTACTS AND LOCATIONS:
Overall Officials: Dio Kavalieratos, PhD, Principal Investigator — Section of Palliative Care and Medical Ethics; Division of General Internal Medicine, University of Pittsburgh; Joseph Pilewski, MD, Principal Investigator — Pulmonary, Allergy, and Critical Care Medicine Division; University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
It is possible that the investigators may use the information obtained from this study in other research studies examining the treatment of Cystic Fibrosis. This information may also be shared with other researchers here and at other research centers, but those researchers will never be provided with any personal identifiers that would allow them to learn participant's identity.